CLINICAL TRIAL: NCT00187785
Title: Doctor-Patient Communication in Spanish
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: UMC200552
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2006-01-18 (Estimated); Status verified 2005-08

CONDITIONS: Upper Respiratory Infection; Hypertension; Diabetes
Keywords: Hispanic; communication
MeSH Terms: conditions — Respiratory Tract Infections; Hypertension; Diabetes Mellitus; Communication

INTERVENTIONS:
Behavioral: Spanish speaker level

SUMMARY:
Does use of a translator or use of less than perfect Spanish diminish provider-patient communication compared to a native speaker.

DETAILED DESCRIPTION:
Spanish speaking drop-in patients will be consented then randomized to receive care by a native Spanish speaker, an English speaker using a translator, or an English speaker with intermediate Spanish skills using Spanish. After the visit, the researcher will enquire about patient satisfaction, when the next appointment is, whether medication has been changed, and what instructions their provider gave them. Each provider will do a similar questionnaire. A blinded researcher will score a concordance of plans between provider and patient to see if there is a significant difference in retained information between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaker

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-09; Study Completion 2006-12

PRIMARY OUTCOMES:
retention of medical information

SECONDARY OUTCOMES:
patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Roger B Mortimer, MD, Principal Investigator — Department of Family Practice
Locations (1):
- UMC Family Health Center, Fresno, California, United States